CLINICAL TRIAL: NCT04996316
Title: Implementing USPSTF Recommendations for Breast Cancer Screening and Prevention by Integrating Clinical Decision Support Tools With the Electronic Health Record
Brief Title: MammoScreen Breast Cancer Risk Assessment and Decision Aid for Breast Cancer Screening and Referrals
Status: Enrolling by invitation | Type: Observational
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Karen Eden, Ph.D., Principal Investigator, OHSU Knight Cancer Institute
Other Study IDs: STUDY00022698; NCI-2021-06583 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00022698 (Other: OHSU Knight Cancer Institute); R01HS027796 (AHRQ)
Record Dates: First submitted 2021-08-02; First posted 2021-08-09 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Interviews as Topic; Educational Status

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

GROUPS / COHORTS (2):
- Clinical staff (interview, training, survey): Before implementation, some participants will complete usability testing of the interface in the electronic health record and MammoScreen. Participants undergo training sessions over 20 minutes and participate in interviews over 30 minutes at baseline, prior to MammoScreen launch. Clinical staff also participate in interviews over 30 minutes after MammoScreen launch during years 2-4. Participants complete surveys during the maintenance phase, about six months after the last reminders are sent.
  Interventions: Other: Electronic Health Record Review; Other: Interview; Other: Survey Administration; Other: Training and Education
- Patients (interview, MammoScreen): Patients participate in interviews up to 1 hour. Patients medical records are reviewed. Patients use the MammoScreen at enrollment. Some Patients will also participate in interviews up to 1 hour, each during years 3-5.
  Interventions: Other: Electronic Health Record Review; Other: Interview; Other: Media Intervention

INTERVENTIONS:
Other: Electronic Health Record Review — Health record reviewed
Other: Interview — Participate in interview
Other: Media Intervention — Use MammoScreen
  Groups: Patients (interview, MammoScreen)
Other: Survey Administration — Complete survey
  Groups: Clinical staff (interview, training, survey)
Other: Training and Education — Undergo training
  Groups: Clinical staff (interview, training, survey)

SUMMARY:
This study collects information to implement MammoScreen for Breast Cancer Screening and Referrals. MammoScreen is a risk assessment questionnaire that identifies individuals at average and increased risk for breast cancer and guides their screening decisions.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Uptake of MammoScreen (the proportion of women who enroll and use MammoScreen, also referred to as Reach.

II. Identification of women with above-average risk for breast cancer by MammoScreen integrated with the electronic health record (EHR).

SECONDARY OUTCOMES:

I. Rates of mammography screening referral. II. Screening completed and mammography results stratified by risk category. III. Among those who meet criteria, genetic counseling referral, visit completed and genetic test done.

OUTLINE:

CLINICAL STAFF: During development some clinical team members will participate in usability testing (up to 30 minutes) of the electronic health record interface with MammoScreen. Some participants will undergo training sessions of about 20 minutes, then participate in interviews lasting up to 30 minutes at baseline prior to MammoScreen launch. Clinical staff also participate in interviews up to 30 minutes after MammoScreen launch during years 2-4. Participants complete surveys during the maintenance phase about six months after the last reminders are sent.

PATIENTS: Patients (enrolled from OHSU IMC) participate in interviews lasting up to 1 hour. Patients medical records are reviewed. Patients will be invited via MyChart to use the MammoScreen. Reminders will be sent via MyChart to non-respondents at 2 and 4 weeks. Patients will use MammoScreen one time right after enrollment. Some patients may also participate in interviews up to 1 hour each during years 3-5.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 40 and 74
* Enrolled in MyChart
* Able to read English

Exclusion Criteria:

* Personal history of breast or ovarian cancer
* Currently Pregnant
* Currently in Hospice

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women between the ages of 40 and 74
Sampling Method: Non-Probability Sample
Enrollment: 1141 (Estimated)
Dates: Start 2022-09-07 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Uptake of MammoScreen | Up to 5 years
  Defined as the proportion of women who enroll and use MammoScreen. Proportions of invitations for newly eligible women and uptake of MammoScreen during the maintenance period, overall and by clinical team, will be characterized along with 95% exact confidence intervals.
Number of women with above-average risk for breast cancer identified by MammoScreen integrated with the electronic health record | Up to 5 years

SECONDARY OUTCOMES:
Rates of mammography screening referral | Up to 5 years
Screening completed | Up to 5 years
  The proportions of patients who open, and complete MammoScreen and 95% confidence intervals will be calculated. Demographic and clinical characteristics of patients who complete MammoScreen versus those who do not will be compared using a two-sample t-test or chi-square test as appropriate. Variation in completing MammoScreen by patient (e.g., age) and provider characteristics (e.g., panel size) will be explored.
Mammography results | Up to 5 years
  Will be stratified by risk category. Will be analyzed similarly using proportions and 95% confidence intervals, and a regression model if allowed by data.
Number of above average risk MammoScreen users who received a genetic counseling referral | Up to 5 years
  Will be analyzed similarly using proportions and 95% confidence intervals, and a regression model if allowed by data.
Number of above average risk MammoScreen users who completed a genetic counseling visit | Up to 5 years
Number of above average risk MammoScreen users who had a genetic test done | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Karen Eden, Ph.D., Principal Investigator — Department of Medical Informatics and Clinical Epidemiology, OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States